CLINICAL TRIAL: NCT06595394
Title: Investigation of the Effect of Exercise Training in Patient With Sarcopenic Multiple Sclerosis
Brief Title: Effect of Combined Exercise Training in Patients With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, tuba kolaylı, Lecturer, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sarcopenicms11
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
Keywords: Sarcopenia; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Sarcopenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Participants were given combined exercise training 3 days a week.
  Interventions: Other: Exercise
- Control group (Active Comparator): Participants were followed with a home program 3 days a week.
  Interventions: Other: Home program

INTERVENTIONS:
Other: Exercise — Participants in the experimental group will receive treatment for 8 weeks, 3 sessions per week. Each treatment session will be planned to last 60 minutes. People in the experimental group will receive a combined exercise training consisting of aerobic exercise, balance exercise and strengthening exercises for 8 weeks.
  Arms: Interventional group
Other: Home program — The control group will be followed with a home program for 8 weeks. Patients will be asked to apply the home program, which includes traditional physiotherapy practices, 3 days a week and this will be followed by physiotherapists.
  Arms: Control group

SUMMARY:
The aim of this clinical trial is exercise in sarcopenic MS patients to demonstrate the effectiveness of education. The main questions it aims to answer are: -Can exercise training make a change in muscle thickness in sarcopenic MS patients?

--Does exercise training have an effect on balance in sarcopenic MS patients?

- Does exercise training have an effect on the risk of falling in sarcopenic MS patients?

Participants will:

They will continue combined exercise applications 3 days a week for 8 weeks. Evaluations will be made before the application and at the end of the 8 weeks. The data will be analyzed afterwards.

DETAILED DESCRIPTION:
A significant decrease in physical performance is observed in MS patients. The reasons for this can be changes in muscle contractile structures and symptoms such as sarcopenia. Sarcopenia is a disorder characterized by loss of skeletal muscle mass and decrease in muscle strength and physical performance. Loss of muscle mass seen outside of old age is defined as secondary sarcopenia. In recent years, studies on neurological disorders and their relationship with sarcopenia have increased. Early diagnosis of sarcopenia in neurological patients and implementation of applications aimed at this are important from an early stage. The aim of this study is to examine the effect of exercise training in sarcopenic MS patients. In the study, participants will be applied a combined exercise program 3 days a week for 8 weeks. Parameters such as muscle thickness, balance, and fall risk will be evaluated before and after physiotherapy application including aerobic exercise, balance exercises, and strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with MS by a neurologist
* People with ambulation whose EDSS is 4.5 or below
* People between the ages of 18-50
* People who do not exercise regularly and are not included in an exercise program

Exclusion Criteria:

* Having been diagnosed with sarcopenia before MS diagnosis
* Having had an MS attack within the last 30 days
* Having any musculoskeletal problems that may affect walking and balance
* Having a diagnosed psychiatric disease that may affect cognitive status
* Having a neurological disease other than MS

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | 8 weeks
  Ultrasound (US) is an easy-to-use imaging method that provides information about both muscle quality and quantity, with no risk of radiation. Muscle thickness will be assessed with US. Muscle thickness assessed with US has been shown to be consistent with gold standard measurements that assess muscle function and thickness.

SECONDARY OUTCOMES:
SARC -F | 8 weeks
  The SARC-F questionnaire was developed in 2018 for the rapid diagnosis of sarcopenia and the questionnaire was recommended in the EWGSOP2 guide in 2019 to determine possible sarcopenia. According to the EWGSOP2 guide, a score of 4 or more (0-10) from the SARC-F questionnaire is considered significant for sarcopenia.
Hand grip strength measurement | 8 weeks
  Muscle strength assessment, which is one of the indicators of sarcopenia, is done by measuring handgrip strength. The measurement is performed with the JAMAR hand dynamometer upon the recommendation of the American Hand Therapists Association. The current cut-off value of handgrip strength is determined as 17.1 kg for men and 11.9 kg for women.
Bioelectrical impedance analysis | 8 weeks
  Bioelectrical impedance analysis (BIA) device is used to determine body composition. At the end of the measurements, if the appendicular skeletal muscle mass is <15 in women and <20 in men according to the cut-off values recommended by EWGSOP2 (European Working Group on Sarcopenia in Older People), this indicates sarcopenia.
Timed Up and Go (TUG) | 8 weeks
  TUG evaluates the functional mobility of patients with the risk of falling. The time it takes for the patient to complete a task is determined with the help of a stopwatch. TUG is an effective and reliable measurement method for the evaluation of functional mobility in patients with MS.
Berg Balance Scale (BBS) | 8 weeks
  BBS was created to assess balance and fall risk. Each question is scored between 0-4 on the 14-item scale. The lowest value obtained from the scale is '0' and the highest value is '56'. According to the total values obtained from the scale; the 0-20 value range indicates severe balance disorder, the 21-40 value range indicates acceptable balance disorder and the 41-56 value range indicates that the patient has good balance.
Fatigue Severity Scale (FSS) | 8 weeks
  The scale consists of 9 questions that allow MS patients to evaluate their last week. All questions are scored between 1-7 and the result is obtained by dividing the total value by 9. A result value greater than 6.1 is a sign of chronic fatigue.
6 Minute Walk Test | 8 weeks
  It is used to evaluate physical performance in people with sarcopenia. The 6MWT can be used safely and easily in the evaluation of impaired functional capacity in outpatient MS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Aksu Yıldırım, Prof., Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No